CLINICAL TRIAL: NCT02031211
Title: Etanercept for the Treatment of Chronic Regional Pain Syndrome
Brief Title: TNF-alpha Inhibition in CRPS: A Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Srinivas Naidu, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29290
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: CRPS; Chronic Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Etanercept; Saline Solution

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Placebo (Placebo Comparator): 0.4 ml/kg of normal saline will be administered subcutaneously.
  Interventions: Drug: Placebo
- Etanercept (Experimental): Patient will receive 0.4 mg/kg of Etanercept subcutaneously twice weekly.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — The patient will receive 0.4 ml/kg as the 25mg/ml preparation subcutaneously.
  Other Names: Enbrel
  Arms: Etanercept
Drug: Placebo — The patient will receive 0.4 ml/kg of Normal Saline injected subcutaneously.
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Studying the effects of Etanercept (an anti-Tumor Necrosis Factor alpha) on early Chronic Regional Pain Syndrome (CRPS). Our hypothesis is that Etanercept will improve patient symptoms if given in early CRPS.

ELIGIBILITY:
Inclusion Criteria:

1. Female pediatric Chronic Regional Pain Syndrome (CRPS) patients with unilateral CRPS of the lower extremity, ages 10-17 years of age.
2. Patients must meet CRPS Type I diagnostic criteria and have current evidence of edema, and a temperature difference between the affected and contralateral limb ≥1.0°C.
3. Duration of symptoms less than 4 months.

Exclusion Criteria:

1. Active malignancy or history of malignancy.
2. Active infection.
3. History of Tuberculosis (TB) or TB exposure.
4. Pregnancy.
5. Concomitant disease causing immunocompromise.
6. Concomitant autoimmune disease such as rheumatoid arthritis, psoriasis, ankylosing spondylitis or Crohn's Disease.
7. Poorly controlled psychiatric disease including anxiety, depression or attention deficit hyperactivity disorder.
8. Hepatic or renal impairment as indicated by serum transaminases and/or creatinine ≥ 150% normal value for age.
9. Evidence of or history of demyelinating disease.

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 8 weeks
  intrapatient comparisons of Visual Analog Scale on Day 35 vs Visual Analog Scale on Day 1, comparing active drug to placebo groups.

SECONDARY OUTCOMES:
Adolescent Pediatric Pain Tool | At end of each week of treatment
  The Adolescent Pediatric Pain Tool is a survey that will be administered at baseline and at the end of each of the four weeks of treatment.
Skin Temperature and Volume of Affected Limb | At beginning and end of study
  The skin temperature and volume of the affected limb will be measured at the beginning and end of the study.
Hospital Anxiety and Depression Scale | Beginning and end of study
  The Hospital Anxiety and Depression Scale is a survey that will be administered at the beginning and end of the study.
Sleep Disturbance Scale for Children | Beginning and end of the study
  The Sleep Disturbance Scale for Children is a survey that will be administered at the beginning and end of the study.
Sleep pattern and quality | Daily
  The patient will sleep with a JawboneUp device, which will measure the sleep pattern and quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States